CLINICAL TRIAL: NCT04475289
Title: Registry for Invasive and Non-invasive Anatomical Assessment and Outcome of Coronary Artery Anomalies
Acronym: NARCO
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00841
Record Dates: First submitted 2020-07-10; First posted 2020-07-17 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Anomalous Coronary Artery Origin; Anomalous Coronary Artery Course; Anomalous Coronary Artery With Aortic Origin and Course Between the Great Arteries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an coronary artery anomaly (focus on ACAOS): Patients eligible for study participation have a CAA and a prior, clinically indicated testing (noninvasive and/or invasive measurement) at our institution to evaluate the hemodynamic significance of this coronary anomaly. They will be approach either after start of this study (retrospective inclusion) or before their testing (prospective inclusion).

SUMMARY:
An anomalous coronary artery from the opposite sinus of Valsalva (ACAOS) represents a congenital disorder with an anomalous location and/or course of the coronary vessel. The prevalence of ACAOS in the general population is around 1 % and they are mostly clinically insignificant and remain often undetected. However, some variants of ACAOS are associated with adverse cardiac events. The possible presence of an interarterial/intramural course is the primary cause for an oval proximal vessel shape and/or proximal vessel narrowing, which may lead under stress conditions to a "dynamic compression" of the vessel (compared to "fixed" stenosis in coronary artery disease). To mimic these conditions, dobutamine and volume challenge is used to invasively measure fractional flow reserve (FFR) during coronary angiography and is seen as the gold standard in assessing the hemodynamic relevance of ACAOS. We established a specialized interdisciplinary clinic for coronary artery anomalies including imaging specialists, invasive cardiologists and congenital heart disease surgeons as correct downstream testing and treatment decision is highly challenging in these patients. Thus, systematic collecting of all available diagnostic methods (invasive and non-invasive) is required to assess the optimal diagnostic procedure and treatment for these patients. Coronary computed tomography angiography (CCTA) is the method of choice to characterize the exact anatomy of ACAOS. However, how functional invasive FFR is associated with anatomical CCTA findings is unknown. Further, diagnostic accuracy of a novel independent research algorithm with computational fluid dynamics (ctFFR) as well as functional imaging (i.e. stress single photon emission computed tomography) in this specific setting is unknown.

The presented project will help to understand the pathophysiology of CAAs with particular focus on ACAOS-IC and improve risk stratification based on non-invasive imaging.

DETAILED DESCRIPTION:
Anomalous coronary arteries (CAA) represent a congenital disorder hallmarked by an anomalous location of the coronary ostium and/or vessel course. Based on the largest study assessing the prevalence and characteristics of CAA detected by coronary computer tomography angiography (CCTA) in Switzerland, the overall prevalence of CAA is 2.6%. However, depending of the type of CAA and its course in relation to the big vessels (aorta and pulmonary artery), not every CAA is accompanied by an increased cardiovascular risk.

Of particular interests are anomalous coronary arteries from the opposite sinus of Valsalva with an interarterial course (ACAOS-IC). Those CAAs represents a congenital disorder with an anomalous location of the coronary ostium and a course of the anomalous vessel between the aorta and the pulmonary artery. The prevalence of ACAOS-IC in the general population is around 1 % and even they are mostly clinically insignificant and remain often undetected.

However, some variants of ACAOS-IC are associated with adverse cardiac events (e.g. sudden cardiac death in young athletes). The possible presence of an intramural course, a course within the aortic wall is the primary cause for an oval proximal vessel shape and proximal vessel narrowing and is suggested to be the primary cause for ischemia. These features may lead under stress conditions to a "dynamic compression" of the vessel (compared to "fixed" stenosis in coronary artery disease). Therefore, to mimic these conditions, dobutamine and volume challenge is used to invasively measure fractional flow reserve (FFRDobutamine) during coronary angiography and is seen as the gold standard in assessing the hemodynamic relevance of ACAOS-IC. Presence of an abnormal FFRDobutamine is one of the most important factors in the decision-making towards surgical repair in ACAOS-IC.

With the frequent use of invasive and non-invasive imaging to rule out coronary artery disease, an increase in absolute numbers of ACAOS-IC is seen and physicians are more confronted with the dilemma of how to manage these patients. Usually the question is whether the ACAOS-IC is a coincidental finding or if the anomaly is causative for the patients' symptoms. Thus, systematic acquisition of all available diagnostic methods (invasive and non-invasive) is required to assess the optimal diagnostic procedure for this patients.

The presented project will help to understand the pathophysiology of CAAs with particular focus on ACAOS-IC and improve risk stratification based on non-invasive imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* CAA with a clinically indicated testing (noninvasive and/or invasive measurement) at our institution
* Informed consent

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients eligible for study participation have a CAA and a prior, clinically indicated testing (noninvasive and/or invasive measurement) at our institution to evaluate the hemodynamic significance of this coronary anomaly.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of revascularization | 5 years
  Frequency of revascularizations (i.e. unroofing, re-implantation of the coronary artery, percutaneous coronary intervention (PCI) and coronary artery bypass graft (CABG) etc.) of the anomalous vessel in patients with CAA.

SECONDARY OUTCOMES:
Quantitative assessment (in SI-Units) of the anatomical features in the coronary computed tomography angiography (CCTA) | 5 years
  The correlation between anatomical features in the CCTA and the primary outcome (frequency of revascularization)
Invasive assessment of hemodynamic relevance | Through clinically indicated diagnostic evaluation, an average of 2 months
  The correlation of invasive assessement under pharmacologic inotropic stress and volume challenge (intravascular ultrasound and fractional flow reserve) with the quantitative determined anatomical features assessed in the CCTA
Computational fluid dynamics | Through clinically indicated diagnostic evaluation, an average of 2 months
  The correlation between FFR-CT and the invasively measured FFR-values
IVUS | Through clinically indicated diagnostic evaluation, an average of 2 months
  The alternation of intravascular ultrasound (IVUS) minimum lumen area at rest and under pharmacologic inotropic stress + volume challenge
Sports | at baseline, one year and 5 year after diagnosis
  Sports behaviour survey

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Gräni, MD PhD, Principal Investigator — Inselspital, Bern University Hospital
Locations (2):
- Switzerland (2):
  - University Hospital Inselspital, Bern, Bern
  - University Hospital, Zürich, Zurich

REFERENCES:
- [Background] Grani C, Buechel RR, Kaufmann PA, Kwong RY. Multimodality Imaging in Individuals With Anomalous Coronary Arteries. JACC Cardiovasc Imaging. 2017 Apr;10(4):471-481. doi: 10.1016/j.jcmg.2017.02.004. PMID 28385257